CLINICAL TRIAL: NCT00665197
Title: Improving Outcomes in Radiotherapy Using New Strategies of Treatment Delivery With Focus on Oesophageal Cancer.
Brief Title: Palliative Radiotherapy and Brachytherapy for Oesophageal Cancer Dysphagia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E3.30.27
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Brachytherapy; Radiotherapy; Palliation; Dysphagia
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Protracted Course Radiotherapy (Active Comparator): High Dose Rate brachytherapy 8.0 Gy x 2
  External beam radiotherapy 30 Gy in 10 fractions of 3.0 Gy
  Interventions: Radiation: Protracted Course Radiotherapy
- Short Course Radiotherapy (Experimental): High Dose Rate brachytherapy 8.0 Gy x 2
  External beam radiotherapy 20 Gy in 5 fractions of 4.0 Gy
  Interventions: Radiation: Short Course Radiotherapy

INTERVENTIONS:
Radiation: Protracted Course Radiotherapy — External Beam Radiation 30 Gy in 10 fractions
  Arms: Protracted Course Radiotherapy
Radiation: Short Course Radiotherapy — External Beam Radiation 20 Gy in 5 fractions
  Arms: Short Course Radiotherapy

SUMMARY:
Hypothesis: In the management of advanced oesophageal cancer, to determine if a shorter regime of external beam radiotherapy (using higher daily doses, and combined with intraluminal high dose rate brachytherapy) is not inferior in the palliation of dysphagia than a more protracted course of external beam radiotherapy (using lower daily doses and combined with equal intraluminal high dose rate brachytherapy).

DETAILED DESCRIPTION:
This is a prospective, pragmatic and multi-centre clinical trial, without blinding or masking to the randomly assigned treatment. Patient registration and randomization are centralized. There are two arms to the study, expecting an equal numbers of patients randomized to each arm. Stratification will by according to: (1) treating institution/country, and (2) baseline Stage (M1 = distant metastases versus M0 = no distant metastases). The primary statistical analysis will be conducted as an "intention-to-treat" clinical trial.

A cost-effectiveness analysis is not required because the main contrast is between 5 and 10 fractions of EBRT, where 5 fractions are less expensive than 10 fractions. This protocol follows the recommendations of CONSORT for the reporting of non-inferiority and equivalence trials. The active control is 30 Gy in 10 fractions, and the new therapy is 20 Gy in 5 fractions.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic and biopsy-proven carcinoma of the esophagus, either Adenocarcinoma or Squamous cell carcinoma;
* Lesions of the thoracic oesophagus and the abdominal oesophagus but not involving the cardia of the stomach. (The oesophagus extends from the cricopharyngeus muscle at the level of the cricoid cartilage to the GEJ junction. The most proximate cervical oesophagus extends approximately 2-3 cm distal to the cricopharyngeus muscle approximately 18 cm from the incisors, and is excluded from this study; however the remaining oesophagus is included in this study, including the last 1-2 cm of the oesophagus which is intra-abdominal and up to the GEJ.);
* Dysphagia immediately prior to the first HDR ILBT session (based on a 4-question summary score of 4-15 (i.e. less than a score of 16) using four of the questions from the EORTC QLQ OES-18 measure;
* Able to insert the intra-esophageal applicator (Dilatation is allowed to open up the tumor/lumen to facilitate insertion, and this does not preclude eligibility. Any oesophageal stent must be removed prior to brachytherapy because metal stents may inappropriately increase the dose of radiation to the esophageal wall by approximately 10%.]);
* Karnofsky is between 40 and 90, inclusive and at baseline (no patient can be 100 as all will have at least dysphagia from disease at baseline; patients with KPS <40 are not eligible for this study);
* Eligible for radiotherapy (e.g. any pacemaker is not within 2.5 cm of the outside of the field edge for the EBRT component of therapy);
* Signed informed consent.

Exclusion Criteria:

* Age less than 18;
* Patients suitable for curative treatment with either surgery or chemo-radiation;
* Tracheo-esophageal fistula, or deep mucosal ulceration;
* Perforation or massive esophageal bleeding ;
* Previous treatment (e.g. chemotherapy, radiation therapy, laser therapy or surgery) for esophageal cancer (gastrostomy or PEG does not constitute exclusion criteria, and should be considered for patients with complete obstruction or where there has been substantial loss in body weight prior to diagnosis);
* Stents in situ (i.e. not removed prior to the first HDR ILBT);
* Previous thoracic radiation therapy for any cause, either EBRT or ILBT;
* Evidence of other uncontrolled malignancies, or evidence of synchronous head and neck or lung primary cancers (regardless of whether those malignancies could be managed with curative intent);
* Failure to complete all baseline assessments required for the study, including patient-elicited scores for symptoms and QOL;
* Pregnant or lactating patients.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Dysphagia relief | 3 years

SECONDARY OUTCOMES:
Quality of life | 3 years
Treatment Toxicity | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Rosenblatt, MD, Study Chair — International Atomic Energy Agency
Locations (7):
- Credit Valley Hospital Statistical Centre, Credit Valley, Ontario, Canada
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China
- University of Zagreb Clinical Hospital, Zagreb, City of Zagreb, Croatia
- Tata Memorial Hospital, Mumbai, Parel, India
- Institute of Nuclear Medicine and Oncology, Lahore, Punjab Province, Pakistan
- University of the Witwatersrand Department of Radiat. Oncology, Johannesburg, Parktown, South Africa
- Mahidol University Faculty of Medicine Siriraj Hospital, Bangkok, Siriraj, Thailand

REFERENCES:
- [Background] Sur RK, Donde B, Levin VC, Mannell A. Fractionated high dose rate intraluminal brachytherapy in palliation of advanced esophageal cancer. Int J Radiat Oncol Biol Phys. 1998 Jan 15;40(2):447-53. doi: 10.1016/s0360-3016(97)00710-4. PMID 9457834
- [Background] Sur RK, Levin CV, Donde B, Sharma V, Miszczyk L, Nag S. Prospective randomized trial of HDR brachytherapy as a sole modality in palliation of advanced esophageal carcinoma--an International Atomic Energy Agency study. Int J Radiat Oncol Biol Phys. 2002 May 1;53(1):127-33. doi: 10.1016/s0360-3016(02)02702-5. PMID 12007950
- [Background] Gaspar LE, Nag S, Herskovic A, Mantravadi R, Speiser B. American Brachytherapy Society (ABS) consensus guidelines for brachytherapy of esophageal cancer. Clinical Research Committee, American Brachytherapy Society, Philadelphia, PA. Int J Radiat Oncol Biol Phys. 1997 Apr 1;38(1):127-32. doi: 10.1016/s0360-3016(97)00231-9. PMID 9212013
- [Background] Kumar MU, Swamy K, Supe SS, Anantha N. Influence of intraluminal brachytherapy dose on complications in the treatment of esophageal cancer. Int J Radiat Oncol Biol Phys. 1993 Dec 1;27(5):1069-72. doi: 10.1016/0360-3016(93)90525-z. PMID 8262829
- See also: IAEA website — http://www.iaea.org